CLINICAL TRIAL: NCT06800781
Title: Prolonged Posterior Pericardial Chest Tube Treatment to Reduce Rates of Postoperative Atrial Fibrillation Following Cardiac Surgery
Brief Title: Prolonged Chest Tube Treatment to Reduce Rates of Atrial Fibrillation Following Cardiac Surgery
Acronym: PROPER
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Region Skane (Other)
Collaborators: The Swedish Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-07117-01
Record Dates: First submitted 2025-01-08; First posted 2025-01-30 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Coronary Arterial Disease (CAD); Valve Replacement; Aortic Surgery
Keywords: Posterior pericardial chest tube; Postoperative atrial fibrillation (POAF)
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control: Standard care (No Intervention): Patients in the control arm will receive 1-2 mediastinal and 0-2 pleural chest tubes (per clinical routine and surgeon's preference). No posterior pericardial chest tube will be inserted in control patients. All other aspects of postoperative care will follow standard clinical routines and will be identical in the intervention and control arms.
- Prolonged treatment with posterior pericardial chest tube plus standard of care (Experimental): All patients will receive chest tubes based on each surgeon's preference. Usually, 1 or 2 tubes are inserted in the mediastinum, and 1 is inserted into each open pleural cavity. Patients in the intervention arm will receive an additional posterior 20Ch chest tube.. In cases where the surgeon routinely inserts 2 mediastinal chest tubes, they will use 1-2 anterior mediastinal tubes in the intervention group, based on their preference. The posterior chest tube will be positioned between the inferior aspect of the heart and the pericardium and connected to an active suction system per routine . Once the remaining chest tubes are extracted, the posterior chest tube will remain positioned in the pericardium and be reconnected from active suction to a collection bag for passive drainage. The chest tube will be removed on postoperative Day 3 or when chest tube output is <50 mL/24 h.
  Interventions: Procedure: Prolonged treatment with posterior pericardial chest tube plus standard care

INTERVENTIONS:
Procedure: Prolonged treatment with posterior pericardial chest tube plus standard care — Prolonged treatment with posterior pericardial chest tube plus standard care All patients will receive chest tubes based on each surgeon's preference. Usually, 1 or 2 tubes are inserted in the mediastinum, and 1 is inserted into each open pleural cavity. Patients in the intervention arm will receive an additional posterior 20Ch chest tube. In cases where the surgeon routinely inserts 2 mediastinal chest tubes, they will use 1-2 anterior mediastinal tubes in the intervention group, based on their preference. The posterior chest tube will be positioned between the inferior aspect of the heart and the pericardium and connected to an active suction system per routine. Once the remaining chest tubes are extracted, the posterior chest tube will remain positioned in the pericardium and be reconnected from active suction to a collection bag for passive drainage. The chest tube will be removed on postoperative Day 3 or when chest tube output is <50 mL/24 h.
  Arms: Prolonged treatment with posterior pericardial chest tube plus standard of care

SUMMARY:
Evacuation of pericardial blood by posterior pericardiotomy or use of a posterior pericardial chest tube lowers postoperative atrial fibrillation (POAF) rates after cardiac surgery by 45-68%. Although it cannot be generalized due to trial undersizing, posterior pericardial chest tube treatment may be a superior alternative to pericardiotomy, given its low risk of procedural complications.

This interventional multicenter trial will assess whether prolonged treatment with a posterior pericardial chest tube lowers POAF rates after cardiac surgery. Investigators will randomize 624 patients undergoing routine cardiac surgery at Nordic sites 1:1 to receive a posterior pericardial chest tube as adjunct to standard care for up to 3 postoperative days or standard care alone. The primary outcome is the proportion of patients with POAF up to 7 days post-surgery; the study will be powered to detect a relative risk reduction of 30% in the intervention arm. Secondary outcomes are AF burden; days with chest tubes and their output; proportion of patients with POAF up to 14 days post-surgery; direct current conversions during hospital admission; length of ICU/hospital stay; postoperative complications, mortality, ischemic stroke, and major bleeding at 30/90 days and 1/3/5 years; and quality of life/postoperative recovery at 90 days and 1 year. This trial may provide quality clinical evidence supporting the adoption of a simple method to prevent POAF, thus reducing healthcare costs.

DETAILED DESCRIPTION:
Postoperative atrial fibrillation (POAF) occurs in 20-50% of cardiac surgery patients and is associated with poorer surgical outcomes. Buildup of fluid in the pericardium due to intraoperative or postoperative bleeding may induce inflammation in the atrial myocardium, leading to POAF. Evacuation of pericardial blood by creating an opening in the pericardium (posterior pericardiotomy) significantly lowers POAF rates after cardiac surgery. However, its clinical use is limited due to several risks, including injury to the pulmonary veins, esophagus, and phrenic nerve. A posterior pericardial chest tube, used routinely by some cardiothoracic surgeons, may be a superior alternative given its low risk of procedural complications.

The PROPER trial is a new Nordic collaboration aiming to evaluate the effect of prolonged posterior pericardial chest tube treatment rates of POAF after cardiac surgery in a randomized, controlled, interventional multicenter trial. The evidence provided by this study will enable direct clinical implementation of the intervention following completion of the trial.

Cardiac surgery results in a local and general inflammatory state, and activation of the autonomic nervous system. These conditions may lead to new-onset POAF. POAF occurs in 20-50% of patients following cardiac surgery and is associated with poorer surgical outcomes, including increased risk of stroke, acute kidney injury, prolonged length of hospital stay, and higher mortality rates. In addition, oral anticoagulation (OAC) treatment is frequently initiated after POAF and is rarely discontinued despite most patients regaining sinus rhythm before hospital discharge and over 90% within 60 days of surgery. OAC treatment exposes the patients to a significant risk of major bleeding complications.

Reports suggest that intraoperative and postoperative bleeding is a significant trigger of POAF through its induction of oxidative stress and inflammation of the atrial myocardium. To this end, several studies have shown that drainage of pericardial blood significantly reduces POAF rates after cardiac surgery. Two meta-analyses suggest that a procedure known as posterior pericardiotomy, which involves making a longitudinal incision in the posterior pericardium, may reduce POAF rates by 55-58%. Most recently, a clinical trial including 420 patients who were randomized to posterior pericardiotomy versus conventional treatment found a 45% lower rate of POAF in the intervention group. Despite the compelling evidence that posterior pericardiotomy reduces the rate of POAF, it is rarely used clinically, likely due to the risk of injuring the pulmonary veins, esophagus, or the phrenic nerve during the procedure. Alternatively, aortic surgery patients who received a posterior pericardial chest tube - which may be a superior alternative due to its low rate of complications - were found to have a 68% lower rate of POAF than patients in the control group. This study, however, was limited by its single-center design, small study sample, and lack of generalizability to other types of cardiac surgery. Whether posterior pericardial chest tubes are a feasible treatment to prevent POAF in surgical patients is still unknown.

The preliminary results demonstrate the feasibility of the planned study to administer posterior pericardial chest tube treatment to cardiac surgery patients and monitor them for arrhythmias using the SmartCardia heart rate monitor. The SmartCardia heart monitor is portable and allows for monitoring of the heart rhythm up to 14 days.

In 2023, investigators in Lund conducted an internal pilot study where 14 patients received either a 20Ch or 18Ch posterior pericardial chest tube with a bellow drain (n=7 in each group). Both chest tubes extracted 150-200 mL blood with no reported physical discomfort; 1 and 3 patients in these arms developed POAF, respectively. As a follow-up to this study, from June to August 2024, investigators treated an additional 8 patients with 20Ch chest tubes and 11 patients with the 18Ch chest tubes to determine which chest tube was best suited for the trial. The 20Ch chest tubes were typically extracted on postoperative day (POD) 3 (IQR 3-3) with a median chest tube output between POD 1 and extraction of 100 (50-125) ml. The 18Ch chest tubes were extracted on POD 3 (IQR 3-3) and evacuated 185 (140-250) ml of fluid between POD 1 and extraction. Patients receiving the 20Ch chest tubes reported a discomfort level of 0.5 (0-1.5) on a visual analog scale (VAS), while those receiving the 18Ch chest tubes reported a level of 0 (0-1). Three patients in the 20Ch group (38%) and 4 patients in the 18Ch group (36%) developed POAF.

Pilot studies have shown that both the 18Ch and the 20Ch chest tubes effectively evacuate blood from the pericardium. Although the 18Ch chest tube evacuated a higher fluid volume on POD 1, upon inspection, no tubes were obstructed by clots after removal. This suggests that the 20Ch chest tube evacuated posterior pericardial blood more efficiently on POD 0 (while connected to the remaining standard tubes), leaving less fluid to be drained on POD 1 and onward. Since nurses at the ward and ICU were more positive towards handling the familiar 20Ch chest tube, and since the manufacturer of the 18Ch chest tubes ran out of stock during the pilot study period, investigators believe that the 20Ch chest tube is the superior alternative for this study.

While no conclusions regarding changes in POAF rates could be drawn from the pilot studies due to the small sample sizes, internal team has in parallel conducted a retrospective, observational study in Iceland on the effect of posterior pericardial chest tube on POAF rates after routine cardiac surgery. Investigators have found that a posterior pericardial chest tube significantly reduced POAF rates in a propensity score-matched population of 1,106 patients undergoing coronary artery bypass grafting and aortic valve replacement (OR 0.66 [95%CI 0.51-0.86], p=0.002). A manuscript detailing the results of this study is currently under revision at The Journal of Cardiothoracic and Vascular Surgery Open.

The current evidence is insufficient to support placing an additional chest tube or to justify its adoption into clinical practice.

Therefore, a large, high-quality, multicenter clinical trial on the effect of posterior pericardial chest tube treatment after cardiac surgery is warranted. The aim of this study is to evaluate whether prolonged treatment with a posterior pericardial chest tube reduces the frequency of POAF after routine cardiac surgery. The SmartCardia monitor will aid in determine whether a patient has experienced POAF during the first 14 postoperative days. If successful, the trial could benefit cardiac surgery patients by reducing the incidence of a disabling postsurgical complication, thereby minimizing patient harm and potentially lowering healthcare costs.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Undergoing non-emergent surgery (>24 hours between decision to operate and surgical procedure) with coronary artery bypass grafting, aortic valve replacement, aortic surgery without the use of circulatory arrest, or any combination of these procedures
* Able to give written informed consent

Exclusion Criteria:

* History of atrial fibrillation (AF) or atrial flutter
* History of electrophysiological interventions or treatment with antiarrhythmic drugs due to arrhythmias other than AF
* Pre- or postoperative prophylactic treatment with amiodarone
* Existing pacemaker, ICD, or CRT device without a functional atrial lead
* Aortic surgery with hypothermic circulatory arrest
* Previous cardiac surgery
* Previous radiation of the chest due to malignancy
* Ongoing infection at time of surgery
* Ongoing treatment with immunosuppressants, including oral corticosteroids
* Patient already included in another interventional clinical trial
* Patient listed abroad, which would render them to be lost to follow-up after discharge
* Patient does not understand study information given in the local language or, for other reasons, is deemed unfit to participate according to the investigators.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 624 (Estimated)
Dates: Start 2025-02-10 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients with POAF the first 7 postoperative days | From enrollment (randomization) to postoperative day 7
  The primary endpoint will be defined as the proportion of patients with POAF (an episode of atrial fibrillation (AF) or atrial flutter sustained for >30 seconds) registred by any available source in the first 7 postoperative days (i.e 12-lead EKG, telemetric monitoring, SmartCardia monitor)

SECONDARY OUTCOMES:
Proportion of patients with POAF until day 14 postoperative | From enrollment to postoperative day 14
  Proportion of patients with POAF during the recording period (defined as the first 14 postoperative days or battery life of the monitor, whichever is first)
Percentage of POAF burden | From application of SmartCardia monitor until end of recording ((defined as the first 14 postoperative days or battery life of the monitor, whichever is first)
  Percentage of time with POAF (POAF burden) during the whole recording period.
Proportion of patients with and frequency of DC conversions during hospital admission | From enrollment to end of hospital stay or until follow up at postoperative day 30 whichever is first
Cumulative dose of amiodarone administered during hospital admission | From enrollment to end of hospital stay or until follow up at postoperative day 30 whichever is first
Length of ICU and hospital stay | From enrollment to end of hospital stay or until follow up at postoperative day 30 whichever is first
Proportion of patients with pericardial tamponade | From enrollment to end of hospital stay or until follow up at postoperative day 30 whichever is first
Proportion of patients requiring re-exploration for bleeding | From enrollment to end of hospital stay or until follow up at postoperative day 30 whichever is first
Proportion of patients with circulatory arrest | From enrollment to end of hospital stay or until follow up at postoperative day 30 whichever is first
Proportion of patients with surgical site infection | From end of surgery to until 1 year follow up
  Until hospital discharge, follow up at 30d, 90d and 1y
Proportion of patients with mediastinitis | From end of surgery to until 1 year follow up
  Until hospital discharge, follow up at 30d, 90d and 1y
Cardiac- or vein graft injury | From enrollment to end of hospital stay or until follow up at postoperative day 30 whichever is first
Proportion of patients receiving OAC treatment | From end of surgery to until 1 year follow up
  Follow up after discharge at 90d and 1y
Proportion of patients requiring pleural drainage | From enrollment to end of hospital stay or until follow up at postoperative day 30 whichever is first
Number of days with a posterior pericardial chest tube | From day of surgery to end of treatment or until follow up at postoperative day 30 whichever is first
Volume of posterior pericardial chest tube output at extraction | From enrollment to end of hospital stay or until follow up at postoperative day 30 whichever is first
Proportion of patients with AF at any time since last assessment | After hospital discharge until 1 year follow up
  Verified by patient report, hospital admission, DC conversion, or electrocardiogram [ECG]) Follow up after discharge at 30d, 90d & 1y
Mortality | After hospital discharge until 5 year follow up
  Data from national health registry Follow up after discharge at 30d, 90d, 1y, 3y & 5y
Proportion of patients with ischemic stroke | From hospital discharge until 5 year follow up
  Follow up after discharge at 30d, 90d, 1y, 3y & 5y
Proportion of patients hospitalized due to bleeding. | From hospital discharge until 5 year follow up
  Follow up after discharge at 30d, 90d, 1y, 3y & 5y
Quality of life survey | From hospital discharge until 1 year follow up
  12-item Short Form Survey Instrument At hospital admisssion, postoperative 90d & 1y
Postoperative recovery | From hospital discharge until 1 year follow up
  Satisfaction with Life scale Follow up postoperative 90d & 1y
Healthcare cost-benefit analysis | From hospital discharge until 5 year follow up
  Follow up at postoperative day 90, 1y, 3y & 5y

CONTACTS AND LOCATIONS:
Overall Officials: Igor Zindovic Zindovic, MD, PhD, Principal Investigator — Region Skåne
Locations (1):
- Lund University hospital, Lund, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sezai, A. et al. Ann Thorac Cardiovasc Surg 27, 191-199, (2021).
- [Background] Rabelo, L. G. et al. Abstract presented at 104th Annual Meeting of AATS, (2024).
- [Background] Fragão-Marques, M. et al. Ann Thorac Cardiovasc Surg 26, 342-351, (2020).
- [Background] Eryilmaz S, Emiroglu O, Eyileten Z, Akar R, Yazicioglu L, Tasoz R, Kaya B, Uysalel A, Ucanok K, Corapcioglu T, Ozyurda U. Effect of posterior pericardial drainage on the incidence of pericardial effusion after ascending aortic surgery. J Thorac Cardiovasc Surg. 2006 Jul;132(1):27-31. doi: 10.1016/j.jtcvs.2006.01.049. PMID 16798298
- [Background] Gillinov, A. M. et al. N Engl J Med 374, 1911-1921, (2016).
- [Background] Kiviniemi, T. et al. Am Heart J 237, 127-134, (2021).
- [Background] Hogue CW Jr, Domitrovich PP, Stein PK, Despotis GD, Re L, Schuessler RB, Kleiger RE, Rottman JN. RR interval dynamics before atrial fibrillation in patients after coronary artery bypass graft surgery. Circulation. 1998 Aug 4;98(5):429-34. doi: 10.1161/01.cir.98.5.429. PMID 9714093
- [Background] Paparella, D. et al. Eur J Cardiothorac Surg 21, 232-244, (2002).
- [Background] Xiong T, Pu L, Ma YF, Zhu YL, Li H, Cui X, Li YX. Posterior pericardiotomy to prevent new-onset atrial fibrillation after coronary artery bypass grafting: a systematic review and meta-analysis of 10 randomized controlled trials. J Cardiothorac Surg. 2021 Aug 14;16(1):233. doi: 10.1186/s13019-021-01611-x. PMID 34391454
- [Background] Gozdek M, Pawliszak W, Hagner W, Zalewski P, Kowalewski J, Paparella D, Carrel T, Anisimowicz L, Kowalewski M. Systematic review and meta-analysis of randomized controlled trials assessing safety and efficacy of posterior pericardial drainage in patients undergoing heart surgery. J Thorac Cardiovasc Surg. 2017 Apr;153(4):865-875.e12. doi: 10.1016/j.jtcvs.2016.11.057. Epub 2016 Dec 19. PMID 28087110
- [Background] Gaudino M, Sanna T, Ballman KV, Robinson NB, Hameed I, Audisio K, Rahouma M, Di Franco A, Soletti GJ, Lau C, Rong LQ, Massetti M, Gillinov M, Ad N, Voisine P, DiMaio JM, Chikwe J, Fremes SE, Crea F, Puskas JD, Girardi L; PALACS Investigators. Posterior left pericardiotomy for the prevention of atrial fibrillation after cardiac surgery: an adaptive, single-centre, single-blind, randomised, controlled trial. Lancet. 2021 Dec 4;398(10316):2075-2083. doi: 10.1016/S0140-6736(21)02490-9. Epub 2021 Nov 14. PMID 34788640
- [Background] St-Onge S, Perrault LP, Demers P, Boyle EM, Gillinov AM, Cox J, Melby S. Pericardial Blood as a Trigger for Postoperative Atrial Fibrillation After Cardiac Surgery. Ann Thorac Surg. 2018 Jan;105(1):321-328. doi: 10.1016/j.athoracsur.2017.07.045. Epub 2017 Nov 24. PMID 29174782
- [Background] Taha A, Nielsen SJ, Bergfeldt L, Ahlsson A, Friberg L, Bjorck S, Franzen S, Jeppsson A. New-Onset Atrial Fibrillation After Coronary Artery Bypass Grafting and Long-Term Outcome: A Population-Based Nationwide Study From the SWEDEHEART Registry. J Am Heart Assoc. 2021 Jan 5;10(1):e017966. doi: 10.1161/JAHA.120.017966. Epub 2020 Nov 30. PMID 33251914
- [Background] Hindricks, G. et al. Eur Heart J 42, 373-498, (2021).
- [Background] El-Chami MF, Kilgo P, Thourani V, Lattouf OM, Delurgio DB, Guyton RA, Leon AR, Puskas JD. New-onset atrial fibrillation predicts long-term mortality after coronary artery bypass graft. J Am Coll Cardiol. 2010 Mar 30;55(13):1370-6. doi: 10.1016/j.jacc.2009.10.058. PMID 20338499